CLINICAL TRIAL: NCT04252963
Title: Double-blind, Randomized, Placebo Controlled, Multicenter, Phase IV Clinical Trial to Assess the Efficacy and Safety of MUCOLASE Tablet (Streptokinase • Streptodornase) in Patients With Acute Upper Respiratory Infection or Acute Bronchitis
Brief Title: Clinical Trial to Assess the Efficacy and Safety of MUCOLASE Tablet(Streptokinase • Streptodornase)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-MUC-401
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Acute Upper Respiratory Infection; Acute Bronchitis
MeSH Terms: conditions — Bronchitis | interventions — Streptodornase and Streptokinase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mucolase (Experimental)
  Interventions: Drug: MUCOLASE tablet (streptokinase • streptodornase)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MUCOLASE tablet (streptokinase • streptodornase) — streptokinase • streptodornase 5mg
  Arms: Mucolase
Drug: Placebo — Placebo of MUCOLASE tablet
  Arms: Placebo

SUMMARY:
A phase 4 study to evaluate efficacy and safety of MUCOLASE tablet (streptokinase • streptodornase)

DETAILED DESCRIPTION:
Double-blind, randomized, placebo controlled, multicenter, phase 4 clinical trial to assess the efficacy and safety of MUCOLASE tablet (streptokinase • streptodornase) in patients with acute upper respiratory infection or acute bronchitis

ELIGIBILITY:
Inclusion Criteria:

* 19≤ age
* Patients with acute upper respiratory infection or acute bronchitis
* Patients with cough and phlegm within 48 hrs as of Visit 1
* Patients understood the consents and purpose of this trial and signed consent form

Exclusion Criteria:

* Patients with high fever (≥39℃)
* Patients with severe respiratory diseases (ex) bronchial asthma, pneumonia, pulmonary tuberculosis, bronchiectasis, mucus sticking, chronic obstructive pulmonary disease (COPD), etc.
* Patients with a history of hypersensitivity to drug
* Patients with abnormal blood coagulation
* Patients with thrombocytopenia
* Patients with uncontrolled hypertension
* Patients with a severe liver disorder(AST or ALT level exceeds 2 times more than normal upper range)
* Patients woth a clinically significant renal failure(MDRD eGFP < 60 mL/min/1.73m2)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in BSS (Bronchitis Severity Score) | baseline, 7 days
  BSS (Bronchitis Severity Score) is derived by summing responses to five major symptoms (i. e. cough, sputum, rales/rhonchi, chest pain during coughing, dyspnoea) with higher scores indicating more severe symptomatology, rated from 0 to 4 (0 = absent, 1 = mild, 2=moderate, 3 = severe, 4 = very severe)

SECONDARY OUTCOMES:
Change from baseline in each symptom score of BSS (Bronchitis Severity Score) | baseline, 7 days
  BSS (Bronchitis Severity Score) is derived by summing responses to five major symptoms (i. e. cough, sputum, rales/rhonchi, chest pain during coughing, dyspnoea) with higher scores indicating more severe symptomatology, rated from 0 to 4 (0 = absent, 1 = mild, 2=moderate, 3 = severe, 4 = very severe)
Change from baseline in cough/sputum domain score of BSS (Bronchitis Severity Score) | baseline, 7 days
  BSS (Bronchitis Severity Score) is derived by summing responses to five major symptoms (i. e. cough, sputum, rales/rhonchi, chest pain during coughing, dyspnoea) with higher scores indicating more severe symptomatology, rated from 0 to 4 (0 = absent, 1 = mild, 2=moderate, 3 = severe, 4 = very severe)
Complete resolution rate of each symptom | 7 days
The number of use of relief drugs | 7 days
Integrative Medicine Outcomes Scale | 7 days
  Integrative Medicine Outcomes Scale is assessed separately by th subjects and thd investigators at end of study, based on BSS of baseline. (Scoring system: 1 = complete recovery, 2 = major improvement, 3 = slight-to-moderate improvement, 4 = no change, 5 =deterioration)
Integrative Medicine Patient Satisfaction Scales | 7 days
  Integrative Medicine Outcomes Scale is assessed by subgects at end of study. (Scoring system: 1 = very satisfied, 2 = satisfied, 3 = neutral, 4 = dissatisfied, 5 =very dissatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Ha Yoo, MD, Ph.D, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea